CLINICAL TRIAL: NCT03038373
Title: Elucidating the Mechanism of Remission of Type 2 Diabetes in Morbid Obese Patients After Bariatric Surgery-focused on Beta Cell Function and Insulin Sensitivity Changes
Brief Title: Elucidating the Mechanism of Remission of Type 2 Diabetes in Morbid Obese Patients After Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dasman Diabetes Institute (Other)
Collaborators: Kuwait University (Other)
Responsible Party: Sponsor
Other Study IDs: RA-2011-014
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2021-10

CONDITIONS: Morbid Obesity; Type2 Diabetes
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, peripheral blood mononuclear cell (PBMC), fat tissues, muscle tissues, remnant surgical tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group I: Morbid Obese Type 2 Diabetics, undergo Laparoscopic Sleeve Gastrectomy
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy
- Group II: Morbid Obese Non Diabetics, undergo Laparoscopic Sleeve Gastrectomy
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy
- Group III: Lean Diabetics, No surgery
- Group IV: Lean Non Diabetics, No surgery

INTERVENTIONS:
Procedure: Laparoscopic Sleeve Gastrectomy — Laparoscopic Sleeve Gastrectomy will be conducted based on standard protocol.
  Groups: Group I; Group II

SUMMARY:
The main aim of this study is to elucidate the mechanism of the remission of type 2 diabetes in the morbid obese patients after laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
In this study four groups including: Group I - Morbid Obese Diabetics, Group II - Morbid Obese Non Diabetics, Group III - Lean Diabetics, and Group IV - Lean Non Diabetics will be studies. The bariatric surgical procedure should include Laparoscopic Sleeve Gastrectomy (LSG). All participants will be assessed by members of a multidisciplinary obesity team including a surgeon, endocrinologist, dietician, and nurse specialist who will usually have input into patient selection.

Briefly the study will be explained to the each participant, and after his/her agreement, the informed Consent Form will be deliver to him/her for completion and signature. Within a week before surgery each enrolled participant of group I and II will be subjected to a medical questionnaire and other routine laboratory analyses before surgery such as fasting glucose, liver, renal, lipid and coagulation profiles. At this time a Mixed Meal Tolerance Test (MMTT) will be performed and blood samples will be collected for further analysis as it is described in the protocol.

Participants in group I and II will be admitted at Dasman Diabetes Institute for post-surgery follow up, performing MMTT, and donating blood samples on days 07, 15, 30, 60, 90, 180, and 360 post-surgery. Adipose, muscle biopsies, and a sample from remnant surgical tissue from these participants will be harvested during of the LSG (days 0). Participants in group I will be asked to monitor their fasting blood glucose level everyday at early morning and the dose of anti-hyperglycemia medications will be adjusted by the recommendation provided by the physician member of team. This data will be recorded as their continuous blood glucose monitoring.

Group III and IV participants, as control groups with no surgical intervention, will be subjected to the medical questionnaire and other routine laboratory analyses and MMTT in just one visit.

All demographic and clinical information collected from the participants will be recorded in the information form identified by identification number (ID number). Only samples from the cases that do not have any post-surgery related complications or not have any emergency clinical condition will be used for genomics and proteomics analysis.

ELIGIBILITY:
Inclusion Criteria:

* adults
* Type 2 diabetes <5 years
* male and female,
* resident of Kuwait,
* who agreed to participate in the study

Exclusion Criteria:

* pregnancy,
* malignancy,
* type 1 diabetes,
* type 2 diabetes with more than 5 years,
* and history with overt heart and/or kidney failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group I and II: eligible candidates will be selected from waiting list of the surgeon, Group III: volunteer lean type 2 diabetics from patient list of Dasman Diabetes Institute Group IV: Invitation to volunteer
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-04; Primary Completion 2022-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinically definition of remission of type 2 diabetes by by fasting blood glucose level < 7.0 mmol and HbA1c <6.5% | 1 year
  Evidence of clinically definition of remission of type 2 diabetes by by fasting blood glucose level < 7.0 mmol and HbA1c <6.5%

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Arefanian, PhD, Principal Investigator — Dasman Diabetes Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al Shawaf E, Al-Ozairi E, Al-Asfar F, Mohammad A, Al-Beloushi S, Devarajan S, Al-Mulla F, Abubaker J, Arefanian H. Atherogenic Index of Plasma (AIP) a Tool to Assess Changes in Cardiovascular Disease Risk Post Laparoscopic Sleeve Gastrectomy. J Diabetes Res. 2020 Aug 1;2020:2091341. doi: 10.1155/2020/2091341. eCollection 2020. PMID 32832558